CLINICAL TRIAL: NCT02032212
Title: A Randomised, Crossover, Relative Bioavailability Study of Nicotine Delivered by an Electronic Vapour Product, a Nicotine Inhalator and a Conventional Cigarette
Brief Title: A Bioavailability Study of Nicotine Delivered by an Electronic Vapour Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ITG EVP G1 S1
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Subjects use the unflavoured EVP on Day 1, the flavoured EVP on Day 2, the nicotine inhalator on Day 3 and the conventional cigarette on Day 4.
  Interventions: Other: EVP unflavoured; Other: EVP flavoured; Other: Nicotine inhalator; Other: Conventional cigarette
- Sequence 2 (Experimental): Subjects use the flavoured EVP on Day 1, the unflavoured EVP on Day 2, the conventional cigarette on Day 3 and the nicotine inhalator on Day 4.
  Interventions: Other: EVP unflavoured; Other: EVP flavoured; Other: Nicotine inhalator; Other: Conventional cigarette
- Sequence 3 (Experimental): Subjects use the nicotine inhalator on Day 1, the conventional cigarette on Day 2, the unflavoured EVP on Day 3 and the flavoured EVP on Day 4.
  Interventions: Other: EVP unflavoured; Other: EVP flavoured; Other: Nicotine inhalator; Other: Conventional cigarette
- Sequence 4 (Experimental): Subjects use the conventional cigarette on Day 1, the nicotine inhalator on Day 2, the flavoured EVP on Day 3 and the unflavoured EVP on Day 4.
  Interventions: Other: EVP unflavoured; Other: EVP flavoured; Other: Nicotine inhalator; Other: Conventional cigarette

INTERVENTIONS:
Other: EVP unflavoured
Other: EVP flavoured
Other: Nicotine inhalator — 15 mg nicotine Nicorette
Other: Conventional cigarette

SUMMARY:
Electronic Vapour Products (EVPs) are a relatively new class of consumer products that are otherwise known as electronic cigarettes. These may look like conventional cigarettes but do not contain tobacco.

The 'vapour' produced by such devices typically consists of humectants (propylene glycol or glycerol), nicotine, water, and flavours.

This trial is to evaluate the pharmacokinetic profile of an EVP.

DETAILED DESCRIPTION:
The principal part of this study evaluates the nicotine pharmacokinetic profile of conventional cigarettes, a nicotine inhalator, an unflavoured EVP and a flavoured EVP.

A second part investigates the nicotine delivery of an EVP with four different nicotine doses.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-35kg/m2
* Subjects must be established smokers
* Subjects must have smoked five to 30 cigarettes per day for at least one year

Exclusion Criteria:

* Subjects who have used nicotine replacement therapy within 14 days of the screening
* Subjects who have donated blood within 12 months preceding study
* Subjects with relevant illness history
* Subjects positive for hepatitis or HIV
* Subjects with history of drug or alcohol abuse
* Subjects with lung function test or vital signs considered unsuitable
* Subjects who are trying to stop smoking

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Subjects in this arm used the unflavoured EVP on Day 1, the flavoured EVP on Day 2, Nicotine inhalator on Day 3 and the conventional cigarette on Day 4.
- Sequence 2: Subjects in this arm used the flavoured EVP on Day 1, the unflavoured EVP on Day 2, the conventional cigarette on Day 3 and the nicotine inhalator on Day 4.
- Sequence 3: Subjects in this arm used the nicotine inhalator on Day 1, the conventional cigarette on Day 2, the unflavoured EVP on Day 3 and the flavoured EVP on Day 4.
- Sequence 4: Subjects in this arm used the conventional cigarette on Day 1, the nicotine inhalator on Day 2, the flavoured EVP on Day 3 and the unflavoured EVP on Day 4.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 3: Subjects in this arm used the Nicotine inhalator on Day 1 and the conventional cigarette on Day 2, the unflavoured EVP on Day 3 and the flavoured EVP on Day 4.
- Sequence 4: Subjects in this arm used the conventional cigarette on Day 1, the Nicotine inhalator on Day 2, the flavoured EVP on Day 3, the unflavoured EVP on Day 4.
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Plasma Concentration
Description: Maximum plasma nicotine concentration (Cmax)
Time Frame: 1, 2, 3, 4, 5, 6, 7, 8, 10, 13, 15, 30, 45, 60 minutes, 2, 4, 6, 8, 12 and 21 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- EVP Unflavoured: Unflavoured e-vapour product
- EVP Flavoured: Flavoured e-vapour product
- Nicotine Inhalator: Nicotine inhalator 15mg
- Conventional Cigarette: Conventional cigarette (commercially available)
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/ml | 3.6 (33.9) | 2.5 (41.6) | 2.5 (45.2) | 21.2 (43.1)

2. Primary Outcome: Area Under the Concentration-time Curve for Plasma Nicotine (AUCt)
Time Frame: 1, 2, 3, 4, 5, 6, 7, 8, 10, 13, 15, 30, 45, 60 minutes, 2, 4, 6, 8, 12 and 21 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/ml
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Number analyzed (Participants) | 12 | 12 | 12 | 12
min*ng/ml | 425.3 (31.4) | 277.2 (33.7) | 320.6 (47.6) | 2247.0 (28.6)

3. Secondary Outcome: Exhaled Carbon Monoxide
Description: Measured with a Smokerlyser device
Time Frame: 25 minutes
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Number analyzed (Participants) | 12 | 12 | 12 | 12
ppm | 2.5 (1.0) | 2.2 (0.72) | 2.3 (0.78) | 14.8 (3.86)

4. Secondary Outcome: Nicotine Withdrawal Symptoms
Description: Withdrawal symptoms were evaluated with the Minnesota Nicotine Withdrawal Scale questionnaire, to which only the 15 questions of the subject's part were completed. Subjects had to rate behaviours (e.g. angry, irritable, frustrated, depressed, restless, insomnia) from 0 (none) to 4 (severe). A higher score means more severe withdrawal symptoms. Scores range from a minimum of 0 to a maximum of 60.
Time Frame: 30 minutes after the third product use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | 6.40 (6.52) | 6.80 (7.32) | 7.50 (7.08) | 8.10 (8.93)

5. Secondary Outcome: Nicotine Craving
Description: Craving was assessed with the Brief Questionnaire of Smoking Urges (QSU-Brief). Subject had to rate 10 statements, such as "I have a desire for a cigarette right now", by a number ranging from 1 (strongly disagree) to 7 (strongly agree). Scores can range from a minimum of 0 to a maximum of 70. A higher score means a stronger urge to smoke a cigarette.
Time Frame: 30 minutes after the third product use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | 24.8 (11.5) | 25.0 (12.9) | 25.6 (12.0) | 22.8 (14.2)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | EVP Unflavoured | EVP Flavoured | Nicotine Inhalator | Conventional Cigarette
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 3/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVP Unflavoured (N=12) | EVP Flavoured (N=12) | Nicotine Inhalator (N=12) | Conventional Cigarette (N=12)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 2 (5) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No